CLINICAL TRIAL: NCT05233046
Title: Case Controlled Blind Randomized Study on Impact of Nutrition and Mental Health Counseling With Mindfulness Program on Perceived Wellness, Dietary Practices and Relationship to Food.
Brief Title: Impact of Mindfulness Program on Perceived Wellness, Eating Habits and Relationship to Food
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aspire Nutrition, LLP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NourishCarolina
Record Dates: First submitted 2021-12-21; First posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Diet, Healthy; Food Habits; Mental Fatigue; Mental Stress; Mental Health Issue; Nutrition Poor; Nutrition Disorders; Eating, Compulsive; Eating Behavior; Eating Disorder Weight Fixation; Eating Disorders; Nutrition, Healthy; Dietary Habits
Keywords: diet; nutrition; counseling; mental health; physical health; work; stress
MeSH Terms: conditions — Feeding Behavior; Mental Fatigue; Stress, Psychological; Malnutrition; Nutrition Disorders; Food Addiction; Feeding and Eating Disorders; Psychological Well-Being | interventions — Nutritional Status

STUDY DESIGN:
Intervention Model Description: Couseling sessions provided by RDs and licensed board certified mental health professionals are trained with standard protocol and evaluated individually. Training protocol includes handbook and virtual instruction with motivational interviewing techniques like using open-ended questions.
  Both study and control group a counseled with standard protocol that includes weekly nutrition services and biweekly mental health services. Study group receives counseling sessions combined with Nourish Carolina program. Control group won't be taught mindfulness-based concepts.
  Standardized focus includes all participants are presented essential nutrition concepts. Also, nutrition and mental health mindfulness sessions will be coordinated and will compliment each other. Each week designed so that the mindful based mini-exercises outlined in Nourish Carolina will have the same theme for both nutrition and mental health sessions.
Who Masked: Participant
Masking Description: The participants will know only that they have been selected for a study but not what group they are in or what the study is investigating.
  The administrators of the study will know what clients have been assigned the study and what participants are in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Impact of Nourish Carolina - Control Group (Experimental): Group A - nutrition (one time/week) and mental health counseling (biweekly) for 12 weeks
  Interventions: Behavioral: Nutrition and Mental health counseling
- Impact of Nourish Carolina - Study Group (Experimental): Group B - nutrition ( one time/week) and mental health counseling (biweekly)with Nourish Carolina for 12 weeks
  Interventions: Behavioral: Nutrition and Mental health counseling with Nourish Carolina

INTERVENTIONS:
Behavioral: Nutrition and Mental health counseling — Nutrition and Mental health counseling with a standardized format included in each session
  Arms: Impact of Nourish Carolina - Control Group
Behavioral: Nutrition and Mental health counseling with Nourish Carolina — Nutrition and Mental health counseling with a standardized format included in each session combined with the intervention of a 12 week immersion of mindfulness based program ,Nourish Carolina, on CMS , school district employees. Nourish Carolina inlcudes, detailed lessons and descriptions with a caledar that includes mindful eating tips, activities, meditations recipes and videos. The program has monthly themes of mindfulness,gratitude and giving
  Arms: Impact of Nourish Carolina - Study Group

SUMMARY:
Mindfulness, seemingly a simple concept, research shows that the impact of mindfulness on the overall wellness of an individual can be helpful (5). Research supports that mindfulness leads to reduced stress, enhanced performance, better focus, and improved approach (7). Areas of mindfulnessare mindful eating,movement and meditation. Application of mindfulness tools in these areas can be beneficial to health outcomes and to create a happier more efficient work environment (9).

Mindful eating shows to improve diet quality and attitudes toward food and eating. Individuals better understand physical hunger/fullness cues, improve nutrient density, weight control,digestion,systolic blood pressure, and stress(2). Disordered eating behaviors have also shown to improve(3). Mindless eating, such as eating while being on the phone, driving, or watching television can have the opposite effect and can be linked to more emotional hunger cues.

Combining mindful eating with diet therapy can lead to healthier food choices and a more positive feeling towards eating and body image, reducing stress and improving the overall wellness of an individual (4). Aspire's experience shows that aspects of teacher's wellness is worsening with ,media reporting more and more employees resigning from their positions every day (wccb,2021). Teachers have voiced their need for more support with their wellbeing. As a result, Aspire Nutrition is targeting school employees through a newly developed mindfulness program titled Nourish Carolina. This program will be focused on improving the overall wellness of participants Participants are enrolled in the study for 12 weeks. All participants will have weekly nutritional counseling and bi-weekly mental health counseling. Study group will have nutrition and mental health counseling with mindfulness activities and control group will receive nutrition and mental health sessions without mindfulness activities. There is a program curriculum so that mental health and nutrition mindfulness activities compliment eachother The mindfulness lessons for study group are divided into 6 nutrition and 6 mental health sessions,for 15 minutes during the session. Positive outcomes could include improved workplace performance as a result of enhancing school employees overall wellness and quality of life by reducing stress levels, improving diet quality, and improving mental health.

DETAILED DESCRIPTION:
Introduction:

Mindfulness is the cultivation of tools and skills that help navigate thoughts, emotions, increase awareness, and be present in the moment. Cultivating mindfulness involves practice and patience using exercises that strengthen the ability to focus (7). Among the many benefits are self-control, objectivity, improved focus, mental clarity and emotional intelligence(5). As a tool for overall wellness, mindfulness has been beneficial. Mindfulness, a state of mind,appears to impact health and wellness in a powerful way (1). Researchers have concluded that self-rated perceptions of health are among the most powerful predictors of subsequent health outcomes (8). When combined with a holistic approach, mindfulness can enhance perceived wellness and improve workplace culture(8).

Mindful eating emphasizes awareness of internal and external sensations and emotions. Studies reveal that mindful eating strategies can lead to weight stabilization, improved digestion, stress reduction, improvements with binge eating episodes and disordered eating establishing an overall better relationship with food (2). Interest in mindful eating has grown as a strategy to eat with less distractions and to improve eating behaviors. The current research supports that combining behavioral strategies such as mindfulness training with nutrition education can lead to an improved relationship with food that reduces risk of chronic disease, promotes more food enjoyment and supports a healthy body image(1). Studies show that mindfulness can be an effective tool in the treatment of unfavorable behaviors such as emotional eating and binge eating(3). Mindfulness addresses shame/guilt often associated with disordered eating behaviors through encouraging nonjudgmental attitudes (3). Mindfulness training develops the skills needed for awareness of thoughts and emotions and non-judgemental acceptance (1) as a result, improvement in abilities to cope emotions that impact overall wellbeing.

What is the project about :

Aspire Nutrition provides nutrition and mental health counseling to teachers throughout North Carolina. Many teachers have expressed an interest in more support with their overall wellness. Over 500 teachers have resigned over the past two months and continue to quit (wccb,2021). In addition to the many challenges that schools face, many staff members are voicing a need for more support with individual wellness and improvements in the work place environment. This study will focus on establishment of a standardized wellness program, Nourish Carolina, with aims to improve self reported dietary habits and perceived wellness of school employees including teachers, administrative staff, cafeteria staff and all other employees.

The Nourish Carolina program encompases both nutrition and mental health counseling with an emphasis on recruitment of skills/tools necessary to cultivate mindfulness in each session. Each participant will participate in the study for three months (12 weeks). There will be a treatment group and a control group. The treatment group will receive both virtual nutrition and mental health counseling with 15 minutes of mindfulness work in each session. The control group will receive virtual nutrition and mental health counseling without any mindfulness support. The participants will attend weekly nutrition sessions and biweekly mental health sessions. This project is designed to investigate the outcomes of the combined nutrition and mental health counseling with an application of mindfulness skills compared to a control group that only receives counseling services with no mindfulness training. The nutrition counseling sessions will be provided by registered and licensed dietitians. Mental health counseling sessions will be provided by licensed, board certified mental health professionals. The treatment group will be the only group to receive both nutrition and mental health counseling with professional support of mindfulness adaptations.To ensure participants receive the same experience, the mental health mindfulness lessons and the nutrition mindfulness lessons and activities will be coordinated so that these lessons focus on similar concepts within the scope of mindfulness. Each weekly nutrition session in both the treatment group and the control group will include standard Nutrition Lesson Plans. Examples of educational concepts included in a standard lesson are as follows: dietary variety, meal planning, grocery shopping, label reading, healthy snacking, and macronutrients.

Hypothesis:

Nourish Carolina program and mindfulness practices introduced in mental health and nutrition counseling sessions will benefit participants by enhancing relationship to food, diet quality and mental health(stress levels).

Our Approach:

Nourish Carolina, is a three month mindfulness program designed to support the health and wellness of teachers by providing nutrition and mental health counseling combined with cultivating skills and the development of tools encouraging mindfulness. The program duration is 12 weeks. The concepts within the program focuses on mindfulness, gratitude and giving. Lesson Plans for nutrition (6 lessons) and mental health (6 lessons) services are provided for the practitioners to introduce during counseling sessions with the participants in the study group. Participants in the control group will not receive mindfulness activities unless it is the appropriate clinical alternative that a client requires.

Each participant will participate in the study for three months. There will be a treatment group and a control group. The treatment group will receive both virtual nutrition and mental health counseling with 15 minutes allocated towards development of mindfulness skills and tools included into each session. The control group will receive virtual nutrition and mental health counseling sessions without any mindful-based support. The participants will attend weekly nutrition sessions and biweekly mental health sessions. This project is designed to investigate the outcomes of combined nutrition and mental health counseling with a focused approach towards cultivation of mindful based skills, compared to a control group, in order to study changes in dietary habits and perceived wellness.

Registered dietitians and licensed, board certified mental health professionals will be trained with a standard protocol. The training protocol for all providers will include a protocol handbook and virtual, group instruction. Virtual training will include motivational interviewing with a special emphasis on using open-ended questions. Nutrition Lesson Plans with prompts for motivational interviewing, Mindfulness Activities ( Both Nutrition and Mental Health) and appropriate handouts are all included in the Nourish Carolina Handbook. All providers will have a handbook. Proper use of the format will be evaluated by performance evaluations during the virtual training.

The treatment group and control group will both experience the same standard nutrition protocol with standardized Lesson Plans and appropriate nutrition counseling.The treatment group and the control group will both have mental health counseling.The treatment group will be the only group to receive the immersion of mindfulness based concepts throughout their nutrition and mental health counseling sessions.

Participant Recruiting:

All school staff members that work at elementary, middle and high schools throughout the district will be informed about the study and are eligible for participation.

Participants will be recruited through email, word of mouth, meetings at individual schools, and support of the district itself. Eligible participants will have the opportunity to sign up to participate in the study on Aspire Nutrition's website: https://www.aspire- nutrition.com/. Randomization of participants will be used to allocate group selection.

Participants will be assigned to the treatment or control group based on the order their application was received. For clarification, the first 10 subjects will be assigned to the control group, the next 10 will be assigned to the treatment group, and so on. All participants must sign a mandatory consent form before participating in the study. Each participant will be able to sign the consent forms electronically . All outstanding questions concerning consent forms will be addressed by telephone or by a virtual zoom orientation. All of a participant's questions will be addressed thoroughly and completely before signing the consent forms. In addition, as the study progresses, if a participant has any questions or complaints that a practitioner can't address, contact Cyrilla Purnell, MPH, RD, LDN Email : research@aspire-nutrition.com Phone: (704) 819-0050

There will be 500 participants for each round of the study. There may be 3-5 trials conducted to reach the desired goal of 2000 total participants.Each participant will be required to complete the 12 week program within 3 months. There will be 3-5 study sessions, to complete the allocated study participant goal.Each participant will be given an extra month grace period to cover weeks they were not able to attend.

Program Evaluation:

All communication with participants and information collected will be conducted through a HIPPA compliant platform. Each participant will be informed on the process of the study, and the requirements and their commitment. Each participant will be assessed with a standard initial consultation. During the initial consultation the participant will have the opportunity to discuss and formulate individual goals and share concerns and experiences. A pre and post evaluation will be administered based on accepted indicators of food choices, nutrition knowledge, and perceived wellness.The questionnaires selected are well validated and widely used to collect information.

Aspire Nutrition will use focus groups to help further develop the study. The focus groups will be used to determine the needs of the school community and the problems faced in the workplace and with wellness . As perceptions of wellness are individualized and specific to a population, the focus group will provide insight regarding the specific population being studied and their perceptions of wellness. The focus groups will be held virtually and will host participants throughout the school district. There will be two virtual focus groups.

What we have done:

Aspire Nutrition has actively worked with teachers since June 2021. Throughout the months of counseling sessions, the team has established relationships with school employees revealing a need for increased support for teachers. In response to this need Aspire Nutrition has partnered with Eat Smart, Move More, a resource tool to encourage healthy choices. In addition,since previous clients respond positively to mindfulness education so mindfulness activities are used in sessions, Upon conducting research on mindful eating and the benefits of incorporating mindfulness into therapeutic nutrition and mental health sessions, the investigator developed a 12 week mindfulness program, Nourish Carolina. This investigation studies the outcomes of Nourish Carolina in a meaningful and beneficial way.

ELIGIBILITY:
Inclusion Criteria:

* School staff members - including all grade levels and positions of elementary, middle and high schools of North Carolina
* Must be able to attend virtual sessions scheduled visits.
* Must be 21 years old

Exclusion Criteria:

* Not an school district employee
* Can not attend virtual session scheduled visits
* An individual who would require a LAR

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-02 (Estimated); Primary Completion 2022-05-15 (Estimated); Study Completion 2022-09-15 (Estimated)

PRIMARY OUTCOMES:
Impact on relationship to food from Mindfulness Program, Nourish Carolina - Comparison of study group with Control Group, using IES2 and clinical reports from nutrition sessions | IES2 at end of the study -12 weeks. Standard Clinical Templates in Simple Practice for note taking during session provide subjective and objective observations for nutrition sessions both control and study group.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their relationship with food. IES2 is widely used and accepted measure developed by Tracy L Tylka Ph D. with Ohio State University. Data collected will be measured as a scale for questionnaires. The scoring procedure is outlined at the bottom of the IES2 and is calculated as a whole number. Standard Clinical Templates in Simple Practice for note taking during session provide subjective and objective observations for nutrition sessions both control and study group.
Impact on Percieved Wellness from Mindfulness program , Nourish Carolia - Comparison of Study Group with Control Group using BIS2, RAND36, and Clinical reports from treatment sessions, mental health and nutrition | These measurements are assessed at the end of the study -12 weeks. Weekly nutrition and biweekly mental health notes for nutrition sessions both control and treatment groups
  Body Image Scale-2 (BIS 2)scoring procedure for the BIS2 will be reflected as a relative scale of all the participants. Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.Standard clinical templates recorded and stored in Simple Practice for note taking during session provide subjective and objective observations for nutrition sessions both control and study group in nutrition and mental health sessions

SECONDARY OUTCOMES:
Impact of Mindfulness Program on Meals per day | Assessed at the end of the study -12 weeks.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their
Imact of Mindfulness Program on Snacks per day | Assessed 12 weeks.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their
Impact of Mindfulness Program on Food Choices | Assessed at 12 weeks.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their
Impact of Mindfulness Program on Food Rules | Assessed at 12 weeks.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their
Impact of Mindfulness Program on emotional eating | Assessed at 12 weeks.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their
Impactof Mindfulness Program on body trust | Assessed at 12 weeks.
  Measured using Intuitive Eating Scale - 2 (IES2) to assess individual's change with their
Impact of Mindfulness Program on health rating | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program on exercise frequency | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program on desire to work | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program on feelings of wellbeing | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program onl daiy movement | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program on stress management | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program on anxiety level | Assessed at 12 weeks.
  Perceived wellness is measured by RAND 36 Item Health Survey. The RAND-36 survey is widely accepted and consists of 36 items that assess eight health concepts: physical functioning, role limitations caused by physical health problems, role limitations caused by emotional problems, social functioning, emotional well-being, energy/fatigue, pain, and general health perceptions. Physical and mental health summary scores are also derived from the eight RAND-36 scales. provides information on what a clinically important difference is for the RAND-36 scales, and provides guidance for summarizing the RAND-36 in a single number.
Impact of Mindfulness Program on body image | Assessed 12 weeks.
  BIS2 - scoring procedure for the BIS2 will be reflected as a relative scale of all the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Kaylee Patrick, RD/LDN, Principal Investigator — Aspire Nutrition Owner; Cyrilla E Purnell, MPH, RD, Study Director — Program Management and Development

IPD SHARING:
Plan to Share IPD: Yes
The information will be made available to other researchers on the Aspire Nutrition website and will be presented at the FENCE nutrition conference next year if application is accepted
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be made available October 15, 2022
Access Criteria: All inquries will be allowed access
URL: http://aspire-nutrition.com

REFERENCES:
- [Background] Shapiro SL, Carlson LE, Astin JA, Freedman B. Mechanisms of mindfulness. J Clin Psychol. 2006 Mar;62(3):373-86. doi: 10.1002/jclp.20237. PMID 16385481
- [Background] Adams T, Bezner J, Steinhardt M. The conceptualization and measurement of perceived wellness: integrating balance across and within dimensions. Am J Health Promot. 1997 Jan-Feb;11(3):208-18. doi: 10.4278/0890-1171-11.3.208. PMID 10165100
- [Background] Sharma, Praveen Kumar, and Rajeev Kumra. "Relationship between Mindfulness, Depression, Anxiety and Stress: Mediating Role of Self-Efficacy." Personality and Individual Differences, vol. 186, 2022, p. 111363., https://doi.org/10.1016/j.paid.2021.111363.
- [Background] Sala M, Vanzhula I, Roos CR, Levinson CA. Mindfulness and Eating Disorders: A Network Analysis. Behav Ther. 2022 Mar;53(2):224-239. doi: 10.1016/j.beth.2021.07.002. Epub 2021 Aug 5. PMID 35227400
- [Background] Alamout MM, Rahmanian M, Aghamohammadi V, Mohammadi E, Nasiri K. Effectiveness of mindfulness based cognitive therapy on weight loss, improvement of hypertension and attentional bias to eating cues in overweight people. Int J Nurs Sci. 2019 Dec 27;7(1):35-40. doi: 10.1016/j.ijnss.2019.12.010. eCollection 2020 Jan 10. PMID 32099857
- [Background] Wilson RE, Marshall RD, Murakami JM, Latner JD. Brief non-dieting intervention increases intuitive eating and reduces dieting intention, body image dissatisfaction, and anti-fat attitudes: A randomized controlled trial. Appetite. 2020 May 1;148:104556. doi: 10.1016/j.appet.2019.104556. Epub 2020 Jan 1. PMID 31901439
- [Background] Oliver A, Hooper S, Lau R, Hutchinson A. Effect of a multidisciplinary rehabilitation program for patients receiving weight management interventions on eating behaviours and health-related quality of life. Obes Res Clin Pract. 2021 May-Jun;15(3):268-274. doi: 10.1016/j.orcp.2021.03.006. Epub 2021 Mar 15. PMID 33736958
- [Background] Godde JU, Yuan TY, Kakinami L, Cohen TR. Intuitive eating and its association with psychosocial health in adults: A cross-sectional study in a representative Canadian sample. Appetite. 2022 Jan 1;168:105782. doi: 10.1016/j.appet.2021.105782. Epub 2021 Nov 3. PMID 34740711
- [Background] Cancelliere C, Cassidy JD, Ammendolia C, Cote P. Are workplace health promotion programs effective at improving presenteeism in workers? A systematic review and best evidence synthesis of the literature. BMC Public Health. 2011 May 26;11:395. doi: 10.1186/1471-2458-11-395. PMID 21615940
- [Background] Penalvo JL, Sagastume D, Mertens E, Uzhova I, Smith J, Wu JHY, Bishop E, Onopa J, Shi P, Micha R, Mozaffarian D. Effectiveness of workplace wellness programmes for dietary habits, overweight, and cardiometabolic health: a systematic review and meta-analysis. Lancet Public Health. 2021 Sep;6(9):e648-e660. doi: 10.1016/S2468-2667(21)00140-7. PMID 34454642
- See also: Teacher workplace resignation — https://www.wccbcharlotte.com/2021/10/20/teachers-leaving-cms-in-droves/
- See also: Teacher workplace resignation — https://www.wfae.org/education/2021-10-18/staff-shortages-hobble-nc-schools-pandemic-recovery-as-teachers-quit-and-subs-are-scarce